CLINICAL TRIAL: NCT06131177
Title: Comparing Nutritional Interventions in Patients With Alcohol-associated Hepatitis: a Randomized Controlled Trial
Brief Title: Nutritional Interventions in Patients With Alcohol-associated Hepatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Juan-Pablo Arab, MD, Associate Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13698
Record Dates: First submitted 2023-08-16; First posted 2023-11-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients are treated with supplementary protein drink
  Interventions: Dietary Supplement: Nutritional supplement
- SOC (standard of Care) (No Intervention): Patient are provided normal hospital diet or meal

INTERVENTIONS:
Dietary Supplement: Nutritional supplement — Protein supplement
  Arms: Treatment

SUMMARY:
Alcohol-associated hepatitis (AH) is a life-threatening condition with high 90-days mortality (up to 40%) and limited treatment options. Previous studies have shown that decreased nutritional intake (less than 21 kcal/kg/day) is associated to a higher mortality compared to patients with a higher caloric intake. Additionally, it has been suggested that subjects with severe AH, should receive a high-protein diet, however, no specific trials have been carried out to address these questions. Thus, the investigators aim to compare nutritional interventions through a randomized controlled trial to assess if a strategy of peripheral parental nutrition (PPN) plus oral nutritional supplementation (ONS) improves outcomes in patients with severe AH. The investigators will compare standard oral intake, enhanced oral intake with IV fluid supplementation, and PPN plus ONS in patients admitted to hospital with severe AH. These results potentially will help guide practitioners on caloric benchmarks targets for patients with severe AH. This study will also assess specific risks and benefits of different nutritional interventions.

ELIGIBILITY:
Inclusion criteria:

* Adult (>18 years) patients admitted with acute severe AH based clinical diagnosis according to NIAAA criteria
* Excessive alcohol consumption for more than 5 years in a row or interrupted
* No more than 60 days of abstinence before the onset of jaundice
* Bilirubin levels >3 mg/dL (>50 umol/L), AST>50 IU/mL, AST/ALT ratio > 1.5
* Abstinence of other causes of liver disease
* MELD score ≥ 20

Exclusion criteria:

* Age < 18 years
* Pregnancy or lactation.
* Allergy or intolerance to the enhanced oral intake formulation or PPN formulation.
* Expected length of stay less than 48 hours.
* Contraindications to IV fluid or PPN administration (fluid overload, suspected bacteremia).
* Presence of drug-induced liver injury (DILI), ischemic hepatitis, biliary duct obstruction, viral hepatitis, autoimmune hepatitis, or Wilson's disease.
* Extrahepatic neoplasia with a life expectancy of less than 6 months.
* History of severe extrahepatic disease (e.g., chronic kidney failure requiring hemodialysis, severe heart disease (NYHA class ≥3), severe chronic lung disease (class ORO ≥3) that confers a survival of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival (30 days) | 30 days
  30 days mortality (%)

SECONDARY OUTCOMES:
Transplant free survival (90 days) | 90 days
  90 day mortality (%)